CLINICAL TRIAL: NCT01313182
Title: Prevention of Surgical Site Infections: Effectiveness of Nasal Povidone-Iodine
Brief Title: Prevention of Surgical Site Infections: Effectiveness of Nasal Povidone-Iodine and Nasal Mupirocin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: New York University (Other); 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11318
Record Dates: First submitted 2011-02-11; First posted 2011-03-11 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3M Skin and Nasal Antiseptic (Active Comparator): Povidone-iodine solution 5% w/w (0.5% available iodine) USP Patient Preoperative Skin Preparation
  Interventions: Drug: 3M Skin and Nasal Antiseptic
- Bactroban Nasal (Active Comparator): Mupirocin calcium ointment, 2%
  Interventions: Drug: mupirocin calcium ointment, 2%

INTERVENTIONS:
Drug: mupirocin calcium ointment, 2% — Approximately one-half of the ointment from the single-use tube should be applied into 1 nostril and the other half into the other nostril twice daily (morning and evening) for 5 days.
  After application, the nostrils should be closed by pressing together and releasing the sides of the nose repetitively for approximately 1 minute. This will spread the ointment throughout the nares.
  Other Names: Bactroban Nasal
  Arms: Bactroban Nasal
Drug: 3M Skin and Nasal Antiseptic — The solution is applied to for 30 seconds to each nostril twice for a total of 2 minutes. The solution is applied by rotating the applicator around the circumference of the nostril for 15 seconds and then rotating the applicator in the anterior nares for 15 seconds.
  Other Names: 3M Skin and Nasal Antiseptic Povidone-iodine solution
  Arms: 3M Skin and Nasal Antiseptic

SUMMARY:
We hypothesize the application of mupirocin or povidone-iodine to the nares is equally effective in short term Staphylococcus aureus(SA)suppression. Our overall study objective is to measure the rate of deep and superficial Surgical Site Infections (SSIs) after primary hip, knee, shoulder and elbow arthroplasty surgery and primary spinal fusion surgery requiring implantation of prosthetic material, when the patient receives either nasal mupirocin or nasal povidone-iodine prior to surgery.

Secondary study objectives include:

1. Measure hospital length of stay and re-admission rates in the mupirocin and povidone-iodine groups.
2. Measure adverse events related to mupirocin and povidone-iodine.
3. Measure rate of SA resistance to mupirocin.

DETAILED DESCRIPTION:
We hypothesize the application of mupirocin or povidone-iodine to the nares is equally effective in short term Staphylococcus aureus(SA)suppression. Our overall study objective is to measure the rate of deep and superficial Surgical Site Infections (SSIs) after primary hip, knee, shoulder and elbow arthroplasty surgery and primary spinal fusion surgery requiring implantation of prosthetic material, when the patient receives either nasal mupirocin or nasal povidone-iodine prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary arthroplasty or spinal fusion surgery
* Age greater than 18 years

Exclusion Criteria:

* Revision arthroplasty
* Revision spinal fusion surgery
* Primary spine surgery without implantation of prosthetic material
* Allergy to mupirocin
* Allergy to povidone-iodine
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1874 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Phillips, MD, Principal Investigator — NYU Langone Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Result] Phillips M, Rosenberg A, Shopsin B, Cuff G, Skeete F, Foti A, Kraemer K, Inglima K, Press R, Bosco J. Preventing surgical site infections: a randomized, open-label trial of nasal mupirocin ointment and nasal povidone-iodine solution. Infect Control Hosp Epidemiol. 2014 Jul;35(7):826-32. doi: 10.1086/676872. Epub 2014 May 21. PMID 24915210

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only patients receiving surgery were considered Started.
Groups:
- 3M Skin and Nasal Antiseptic: Povidone-iodine solution 5% w/w (0.5% available iodine) USP Patient Preoperative Skin Preparation
  Povidone-iodine solution 5% w/w (0.5% available iodine) Patient Preoperative Skin Preparation: The solution is applied to for 30 seconds to each nostril twice for a total of 2 minutes. The solution is applied by rotating the applicator around the circumference of the nostril for 15 seconds and then rotating the applicator in the anterior nares for 15 seconds.
- Bactroban Nasal: Mupirocin calcium ointment, 2%
  mupirocin calcium ointment, 2%: Approximately one-half of the ointment from the single-use tube should be applied into 1 nostril and the other half into the other nostril twice daily (morning and evening) for 5 days.
  After application, the nostrils should be closed by pressing together and releasing the sides of the nose repetitively for approximately 1 minute. This will spread the ointment throughout the nares.
Period: Overall Study
Arm/Group | 3M Skin and Nasal Antiseptic | Bactroban Nasal
Started | 842 | 855
Completed | 776 | 763
Not Completed | 66 | 92
Not completed — Protocol Violation | 66 | 92

BASELINE CHARACTERISTICS:
Population: arthroplasty or spine fusion surgery patients
Groups:
- Total: Total of all reporting groups
Arm/Group | 3M Skin and Nasal Antiseptic | Bactroban Nasal | Total
Number analyzed (Participants) | 842 | 855 | 1697
Age, Continuous [Mean (Full Range); unit: years] | 61.8 [19.1 to 92.4] | 62.4 [19.2 to 93.2] | 62.1 [19.1 to 93.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 499 | 523 | 1022
  Male | 343 | 332 | 675
Region of Enrollment [Number; unit: participants]
  United States | 842 | 855 | 1697

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Infections Occurring Within 12 Months of Surgical Procedure
Description: Measure the rate (number and percent of patients) with deep and superficial surgical site infections after primary orthopedic surgery and primary spinal fusion surgery requiring implantation of prosthetic material.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | 3M Skin and Nasal Antiseptic | Bactroban Nasal
Number analyzed (Participants) | 776 | 763
participants | 0 | 5

2. Secondary Outcome: Measure Hospital Length of Stay in the Mupirocin and Povidone-iodine Groups.
Description: The hospital length of stay will be measured in the Mupirocin and Povidone-iodine groups.
Time Frame: Post-surgery
Population: Data was not collected for this assessment.
Arm/Group | 3M Skin and Nasal Antiseptic | Bactroban Nasal
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Measure Rate of Staphylococcus Aureus Resistance to Mupirocin.
Description: Lab cultured isolates - they will measure rate of Staphylococcus aureus resistance to mupirocin. Both arms were sampled and tested post-op.
Time Frame: Isolates collected and frozen immediately post-surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | 3M Skin and Nasal Antiseptic | Bactroban Nasal
Number analyzed (Participants) | 842 | 855
Participants | 21 | 24

4. Secondary Outcome: Re-admission Rates in the Mupirocin and Povidone-iodine Groups.
Description: Re-admission rates in the Mupirocin and Povidone-iodine Groups.
Time Frame: 12 months
Population: Data was not collected for this assessment.
Arm/Group | 3M Skin and Nasal Antiseptic | Bactroban Nasal
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | 3M Skin and Nasal Antiseptic | Bactroban Nasal
All-Cause Mortality (participants affected / at risk) | 0/842 | 0/855
Serious Adverse Events (participants affected / at risk) | 0/842 | 0/855
Other Adverse Events (participants affected / at risk) | 15/842 | 76/855
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3M Skin and Nasal Antiseptic (N=842) | Bactroban Nasal (N=855)
Headache (Vascular disorders) | 2 (2) | 15 (15)
Rhinorrhea (General disorders) | 1 (1) | 47 (47)
Nasal irritation (General disorders) | 8 (8) | 13 (13)
Congestion (General disorders) | 3 (3) | 15 (15)
Cough (General disorders) | 3 (3) | 6 (6)
Pharyngeal pain (General disorders) | 0 (0) | 10 (10)

LIMITATIONS AND CAVEATS:
Study failed to achieve target enrollment. The small sample size precluded a multivariate analysis. Nasal culture alone was used as a screen for S. aureus colonization, which has a sensitivity of only 48% to 66%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes